CLINICAL TRIAL: NCT07248228
Title: A Randomized Phase 2 Trial of Memory Avoidance Whole Brain Radiotherapy Versus Hippocampal Avoidance Whole Brain Radiotherapy (Athena 2 Trial)
Brief Title: Memory Avoidance Whole Brain Radiotherapy vs Hippocampal Avoidance Whole Brain Radiotherapy (Athena 2 Trial)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE7325
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Brain Metastases
Keywords: Whole brain radiotherapy; Memory-avoidance whole brain radiotherapy; Hippocampal-avoidance whole brain radiotherapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memory Avoidance Whole Brain Radiation Therapy (MA-WBRT) (Experimental)
  Interventions: Radiation: MA-WBRT (Memory Avoidance Whole Brain Radiation Therapy (MA-WBRT)); Drug: Memantine
- Hippocampal Avoidance Whole Brain Radiation Therapy (HA-WBRT) (Active Comparator)
  Interventions: Radiation: HA-WBRT (Hippocampal Avoidance Whole Brain Radiation Therapy (HA-WBRT)); Drug: Memantine

INTERVENTIONS:
Radiation: MA-WBRT (Memory Avoidance Whole Brain Radiation Therapy (MA-WBRT)) — Participants will receive 10 daily fractions of WBRT per standard of care. Participants receiving MA-WBRT will receive WBRT that avoids the hippocampus, the amygdala, corpus callosum, fornix, hypothalamus, and pituitary.
  Arms: Memory Avoidance Whole Brain Radiation Therapy (MA-WBRT)
Radiation: HA-WBRT (Hippocampal Avoidance Whole Brain Radiation Therapy (HA-WBRT)) — Participants will receive 10 daily fractions of WBRT per standard of care. Participants receiving HA-WBRT will receive WBRT that avoids the hippocampus.
  Arms: Hippocampal Avoidance Whole Brain Radiation Therapy (HA-WBRT)
Drug: Memantine — Memantine is prescribed per standard of care. Participants will continue on memantine for 24 weeks.
  The target dose for memantine is 20 mg (10 mg divided twice daily). Dose is escalated by 5 mg per week to target of 10 mg twice daily (i.e., 5 mg a day for week 1, then 5 mg twice daily for week 2, then 10 mg in the morning and 5 mg in the evening for week 3, then 10 mg in the morning and 10 mg in the evening by week 4).
  Participants will also be prescribed extended release memantine. The target dose for extended release memantine is 28 mg. Dose is escalated by 7 mg per week to target of 28 mg daily (i.e., 7 mg a day for week 1, then 14 mg a day for week 2, then 21 mg a day for week 3, then 28 mg a day for by week 4).

SUMMARY:
Participants in this research study have cancer that has spread to their brain, called brain metastases. One treatment for this type of cancer is called whole brain radiotherapy that stays away from a specific neurocognitive substructure, called the hippocampus, combined with medication to preserve cognitive function. This study compares that approach to another approach of whole brain radiotherapy that stays away from additional structures that are thought to have a role in cognitive function. Researchers want to see if there is a difference in the preservation of cognitive function between these two approaches.

DETAILED DESCRIPTION:
Brain metastases happen when cancer spreads from its original location to the brain. For people with brain metastases, whole brain radiotherapy (WBRT) is important in reducing neurologic symptoms and maximizing intracranial control. Previous studies have shown that adding a drug called memantine to WBRT can help lower the risk of cognitive decline. Previous studies have also shown that hippocampal avoidance WBRT (HA-WBRT) with memantine can reduce the risk of cognitive decline even more. This combination is considered a standard of care option for people with brain metastases.

Even though HA-WBRT successfully reduces the risk of cognitive decline for people with brain metastases, many people still experience some cognitive decline. This means that new treatments are needed to better protect brain function for this population. While avoiding the hippocampus is helpful, there are still many other parts of the brain that may be affected by radiation. Important cognitive structures such as the amygdala, corpus callosum, and fornix are involved with memory processing, executive function, complex task performance, memory formation, and recall. Avoiding these cognitive structures can further preserve cognition for people receiving WBRT.

This study investigates the avoidance of additional cognitive structures (the amygdala, corpus callosum, fornix, hypothalamus, and pituitary) with memory avoidance whole brain radiotherapy (MA-WBRT). The safety and feasibility of MA-WBRT has already been demonstrated. The purpose of this study is to compare MA-WBRT with memantine to HA-WBRT with memantine, which is currently the standard of care for people with extensive brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically, cytologically, or radiographically confirmed diagnosis of solid tumor with brain metastases
* Age >18 years
* Performance status: Karnofsky Performance Status (KPS) ≥ 70
* Estimated life expectancy of at least 3 months
* Participant must be considered a candidate for WBRT by the treating physician
* Participant must be a primary English speaker and have the ability to understand and the willingness to sign an English written informed consent document
* Participant has at least 10 brain metastases or is otherwise suitable for WBRT

Exclusion Criteria:

* Prior whole brain radiation
* Participant has Multiple Sclerosis, Alzheimer's, dementia, or mental disability
* Pregnant or breastfeeding women are excluded from this study.
* Participant is not able to receive an MRI
* Participant has metastasis within avoidance neurocognitive substructures (hippocampus, amygdala, fornix, corpus callosum, pituitary, amygdala)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Time to neurocognitive failure (NCF) | Up to 12 months
  Time to NCF is defined as cognitive decline on the reliable change index (RCI) on at least one of the following tests: HVLT-R, TMT A/B, COWAT, BVMT-R. Tests are defined below.
Hopkins Verbal Learning Test-Revised (HVLT-R) | Day 1 (prior to WBRT treatment)
  The HVLT-R involves three learning trials: Total Recall, Delayed Recall, and Delayed Recognition. The HVLT-R is administered by the examiner reading a 12-item list of words and asking the participant to recall as many as possible (Total Recall). After a 20-25 minutes interval of unrelated tasks, the examiner asks the participant to recall as many words as possible from the original list (Delayed Recall). Then, the examiner reads a 24-item list of words, where 12 words were on the original list and 12 were not (Delayed Recognition). The examiner asks the participant to respond "yes" if the word was on the original list or "no" if it was not. The HVLT-R is scored by summing the number of correctly recalled words across the three trials. Higher scores indicate greater recall.
Hopkins Verbal Learning Test-Revised (HVLT-R) | Month 3
  The HVLT-R involves three learning trials: Total Recall, Delayed Recall, and Delayed Recognition. The HVLT-R is administered by the examiner reading a 12-item list of words and asking the participant to recall as many as possible (Total Recall). After a 20-25 minutes interval of unrelated tasks, the examiner asks the participant to recall as many words as possible from the original list (Delayed Recall). Then, the examiner reads a 24-item list of words, where 12 words were on the original list and 12 were not (Delayed Recognition). The examiner asks the participant to respond "yes" if the word was on the original list or "no" if it was not. The HVLT-R is scored by summing the number of correctly recalled words across the three trials. Higher scores indicate greater recall.
Hopkins Verbal Learning Test-Revised (HVLT-R) | Month 6
  The HVLT-R involves three learning trials: Total Recall, Delayed Recall, and Delayed Recognition. The HVLT-R is administered by the examiner reading a 12-item list of words and asking the participant to recall as many as possible (Total Recall). After a 20-25 minutes interval of unrelated tasks, the examiner asks the participant to recall as many words as possible from the original list (Delayed Recall). Then, the examiner reads a 24-item list of words, where 12 words were on the original list and 12 were not (Delayed Recognition). The examiner asks the participant to respond "yes" if the word was on the original list or "no" if it was not. The HVLT-R is scored by summing the number of correctly recalled words across the three trials. Higher scores indicate greater recall.
Hopkins Verbal Learning Test-Revised (HVLT-R) | Month 9
  The HVLT-R involves three learning trials: Total Recall, Delayed Recall, and Delayed Recognition. The HVLT-R is administered by the examiner reading a 12-item list of words and asking the participant to recall as many as possible (Total Recall). After a 20-25 minutes interval of unrelated tasks, the examiner asks the participant to recall as many words as possible from the original list (Delayed Recall). Then, the examiner reads a 24-item list of words, where 12 words were on the original list and 12 were not (Delayed Recognition). The examiner asks the participant to respond "yes" if the word was on the original list or "no" if it was not. The HVLT-R is scored by summing the number of correctly recalled words across the three trials. Higher scores indicate greater recall.
Hopkins Verbal Learning Test-Revised (HVLT-R) | Month 12
  The HVLT-R involves three learning trials: Total Recall, Delayed Recall, and Delayed Recognition. The HVLT-R is administered by the examiner reading a 12-item list of words and asking the participant to recall as many as possible (Total Recall). After a 20-25 minutes interval of unrelated tasks, the examiner asks the participant to recall as many words as possible from the original list (Delayed Recall). Then, the examiner reads a 24-item list of words, where 12 words were on the original list and 12 were not (Delayed Recognition). The examiner asks the participant to respond "yes" if the word was on the original list or "no" if it was not. The HVLT-R is scored by summing the number of correctly recalled words across the three trials. Higher scores indicate greater recall.
Controlled Oral Word Association Test (COWAT) | Day 1 (prior to WBRT treatment)
  The COWAT is a verbal fluency test that involves the examiner asking the participant to name as many words as they can that start with a designated letter, excluding proper nouns, for one minute. This is repeated three times. The examiner records the words provided by the participant, and the COWAT is scored by calculating the total number of acceptable words that the participant produced. Greater scores indicate a higher performance (greater cognitive capabilities) on the test.
Controlled Oral Word Association Test (COWAT) | Month 3
  The COWAT is a verbal fluency test that involves the examiner asking the participant to name as many words as they can that start with a designated letter, excluding proper nouns, for one minute. This is repeated three times. The examiner records the words provided by the participant, and the COWAT is scored by calculating the total number of acceptable words that the participant produced. Greater scores indicate a higher performance (greater cognitive capabilities) on the test.
Controlled Oral Word Association Test (COWAT) | Month 6
  The COWAT is a verbal fluency test that involves the examiner asking the participant to name as many words as they can that start with a designated letter, excluding proper nouns, for one minute. This is repeated three times. The examiner records the words provided by the participant, and the COWAT is scored by calculating the total number of acceptable words that the participant produced. Greater scores indicate a higher performance (greater cognitive capabilities) on the test.
Controlled Oral Word Association Test (COWAT) | Month 9
  The COWAT is a verbal fluency test that involves the examiner asking the participant to name as many words as they can that start with a designated letter, excluding proper nouns, for one minute. This is repeated three times. The examiner records the words provided by the participant, and the COWAT is scored by calculating the total number of acceptable words that the participant produced. Greater scores indicate a higher performance (greater cognitive capabilities) on the test.
Controlled Oral Word Association Test (COWAT) | Month 12
  The COWAT is a verbal fluency test that involves the examiner asking the participant to name as many words as they can that start with a designated letter, excluding proper nouns, for one minute. This is repeated three times. The examiner records the words provided by the participant, and the COWAT is scored by calculating the total number of acceptable words that the participant produced. Greater scores indicate a higher performance (greater cognitive capabilities) on the test.
Brief Visuospatial Memory Test-Revised (BVMT-R) | Day 1 (prior to WBRT treatment)
  The BVMT-R test involves a participant viewing a page of six figures for 10 seconds and then being asked to draw as many figures as they can remember in their correct places. This is repeated three times. Then, after a 25 minute interval, the examiner asks the participant to recall and draw the figures again. The BVMT-R is scored by summing how many items the participant correctly recalled for each trial. Higher scores indicate higher performance (greater cognitive capabilities) on the test.
Brief Visuospatial Memory Test-Revised (BVMT-R) | Month 3
  The BVMT-R test involves a participant viewing a page of six figures for 10 seconds and then being asked to draw as many figures as they can remember in their correct places. This is repeated three times. Then, after a 25 minute interval, the examiner asks the participant to recall and draw the figures again. The BVMT-R is scored by summing how many items the participant correctly recalled for each trial. Higher scores indicate higher performance (greater cognitive capabilities) on the test.
Brief Visuospatial Memory Test-Revised (BVMT-R) | Month 6
  The BVMT-R test involves a participant viewing a page of six figures for 10 seconds and then being asked to draw as many figures as they can remember in their correct places. This is repeated three times. Then, after a 25 minute interval, the examiner asks the participant to recall and draw the figures again. The BVMT-R is scored by summing how many items the participant correctly recalled for each trial. Higher scores indicate higher performance (greater cognitive capabilities) on the test.
Brief Visuospatial Memory Test-Revised (BVMT-R) | Month 9
  The BVMT-R test involves a participant viewing a page of six figures for 10 seconds and then being asked to draw as many figures as they can remember in their correct places. This is repeated three times. Then, after a 25 minute interval, the examiner asks the participant to recall and draw the figures again. The BVMT-R is scored by summing how many items the participant correctly recalled for each trial. Higher scores indicate higher performance (greater cognitive capabilities) on the test.
Brief Visuospatial Memory Test-Revised (BVMT-R) | Month 12
  The BVMT-R test involves a participant viewing a page of six figures for 10 seconds and then being asked to draw as many figures as they can remember in their correct places. This is repeated three times. Then, after a 25 minute interval, the examiner asks the participant to recall and draw the figures again. The BVMT-R is scored by summing how many items the participant correctly recalled for each trial. Higher scores indicate higher performance (greater cognitive capabilities) on the test.
Trail Making Test (TMT) | Day 1 (prior to WBRT treatment)
  The TMT consists of two parts: Part A and Part B. In Part A, participants are asked to connect 25 circles numbered 1-25 in ascending order. In Part B, participants are asked to connect 13 circles alternating between numbers and letters in ascending order. Participants are asked to complete these tasks as quickly as they can without lifting their pen from the paper. The TMT is measured by the time in seconds that it takes participant to complete the tasks. Higher times indicate greater cognitive impairment.
Trail Making Test (TMT) | Month 3
  The TMT consists of two parts: Part A and Part B. In Part A, participants are asked to connect 25 circles numbered 1-25 in ascending order. In Part B, participants are asked to connect 13 circles alternating between numbers and letters in ascending order. Participants are asked to complete these tasks as quickly as they can without lifting their pen from the paper. The TMT is measured by the time in seconds that it takes participant to complete the tasks. Higher times indicate greater cognitive impairment.
Trail Making Test (TMT) | Month 6
  The TMT consists of two parts: Part A and Part B. In Part A, participants are asked to connect 25 circles numbered 1-25 in ascending order. In Part B, participants are asked to connect 13 circles alternating between numbers and letters in ascending order. Participants are asked to complete these tasks as quickly as they can without lifting their pen from the paper. The TMT is measured by the time in seconds that it takes participant to complete the tasks. Higher times indicate greater cognitive impairment.
Trail Making Test (TMT) | Month 9
  The TMT consists of two parts: Part A and Part B. In Part A, participants are asked to connect 25 circles numbered 1-25 in ascending order. In Part B, participants are asked to connect 13 circles alternating between numbers and letters in ascending order. Participants are asked to complete these tasks as quickly as they can without lifting their pen from the paper. The TMT is measured by the time in seconds that it takes participant to complete the tasks. Higher times indicate greater cognitive impairment.
Trail Making Test (TMT) | Month 12
  The TMT consists of two parts: Part A and Part B. In Part A, participants are asked to connect 25 circles numbered 1-25 in ascending order. In Part B, participants are asked to connect 13 circles alternating between numbers and letters in ascending order. Participants are asked to complete these tasks as quickly as they can without lifting their pen from the paper. The TMT is measured by the time in seconds that it takes participant to complete the tasks. Higher times indicate greater cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Haley Perlow, MD, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Compiled and analyzed participant data will be published upon study completion. Publisher may request Protocol and Statistical Analysis Plan.